CLINICAL TRIAL: NCT07008495
Title: Testicular Sperm Retrieval Rate After Varicocele Ligation in Men With Non Obstructive Azoospermia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Yacoub Nagah Abdelwahab, Resident at Urology Department, Faculty of Medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Non-Obstructive Azoospermia
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-09

CONDITIONS: Non-obstructive Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of varicocele ligation (Active Comparator): About 25 male patients will undergo varicocele ligation then microTESE.
  Interventions: Procedure: varicocelectomy
- Group of TESE (Active Comparator): About 25 male patients will undergo microTESE without varicocele ligation.
  Interventions: Procedure: varicocelectomy

INTERVENTIONS:
Procedure: varicocelectomy — to detect testicular sperm retrieval rate after varicocelectomy in men with non obstructive azoospermia.
  Other Names: TESE

SUMMARY:
A varicocele is an abnormal dilatation and tortuosity of the veins of the spermatic cord. Although varicoceles are common in the general population and are frequently found on routine physical examinations, they represent the most common correctable cause of male factor infertility.

Male factor infertility affects up to half of all couples struggling to conceive, and 10-20% of men evaluated for infertility are found to be azoospermic.

DETAILED DESCRIPTION:
Generally, azoospermia is classified as obstructive azoospermia (OA) or non-obstructive azoospermia (NOA). While OA is obviously caused by obstruction, NOA has many possible causes and is more difficult to manage.

Non-obstructive azoospermia (NOA) is most often a result of primary testicular dysfunction, Varicoceles are found in 20% of the general male population, in up to 40% of men with infertility, and specifically 4.3-13.3% of men with NOA.

The role of varicoceles in NOA has not been fully elucidated. The current best practice statement on the evaluation of azoospermic males from the AUA acknowledges that impaired spermatogenesis associated with varicoceles may be reversible but does not give a clear recommendation for management.

The primary advantage of varicocelectomy in cases of NOA is the possibility of getting motile sperms in the ejaculate. Other benefit of varicocele repairs in azoospermic men is that there are increased success rates of assisted reproductive techniques (ART) such as intracytoplasmic sperm injection (ICSI) or testicular sperm extraction (TESE).

ELIGIBILITY:
Inclusion Criteria:

* Men with non obstructive azoospermia.
* Clinically palpable varicocele ( unilateral or bilateral ).

Exclusion Criteria:

* Known cases of obstructive azoospermia.
* Non palpable varicocele.
* Uncorrectable female causes of infertility.
* genetic abnormalities like klinefelter syndrome.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Sperm retrieval rate | Two Weeks
  Evaluation of Sperm retrieval rate after varicocelectomy in men with non obstructive azoospermia

SECONDARY OUTCOMES:
fertility rate | 3 months from the operation
  Evaluation of fertility rate after varicocelectomy in men with non obstructive azoospermia

CONTACTS AND LOCATIONS:
Overall Officials: Gamal A. Alsagheer, Professor, Study Chair — Urology Department, Faculty of Medicine, South Valley University, Qena, Egypt
Locations (1):
- South Valley University Hospital, Qina, South Valley, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol